CLINICAL TRIAL: NCT05732402
Title: An Open-Label, Multiple-Ascending Dose Study to Assess the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Different Dose Levels of Povetacicept in Subjects With Autoantibody-Associated Glomerular Diseases (RUBY-3)
Brief Title: An Open-label Study of Povetacicept in Autoantibody-Associated Glomerular Diseases
Acronym: RUBY-3
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alpine Immune Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIS-D03
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Lupus Nephritis; Immunoglobulin A Nephropathy; Membranous Nephropathy; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
Keywords: IgA nephropathy; glomerulonephritis, IgA; Immunoglobulin A nephropathy; Berger disease; lupus nephritis; lupus glomerulonephritides; primary membranous nephropathy; membranous nephropathy; glomerulonephritis, membranous; PLA2R; THSD7A; ALPN-303; povetacicept; RUBY-3; RUBY3; Gd-IgA1; GdIgA1; anti-neutrophil cytoplasmic antibody associated vasculitis; ANCA Vasculitis; AAV; Microscopic polyangiitis; Granulomatosis with polyangiitis; Eosinophilic granulomatosis with polyangiitis; Wegener's granulomatosis; Churg-Strauss Disease; Myeloperoxidase (MPO); Proteinase 3 (PR3)
MeSH Terms: conditions — Lupus Nephritis; Glomerulonephritis, IGA; Glomerulonephritis, Membranous; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Microscopic Polyangiitis; Granulomatosis with Polyangiitis; Churg-Strauss Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Povetacicept (Experimental): Part A: Participants will receive povetacicept for 24 weeks with the possibility of participating in treatment extensions through 104 weeks of treatment.
  Part B: Participants with IgAN and pMN will receive povetacicept for an additional 52 weeks.
  Interventions: Drug: Povetacicept

INTERVENTIONS:
Drug: Povetacicept — Administered by subcutaneous injection every 4 weeks
  Other Names: ALPN-303

SUMMARY:
The goal of this clinical study is to evaluate multiple dose levels of povetacicept in adults with immunoglobulin A (IgA) nephropathy (IgAN), primary membranous nephropathy (pMN), lupus-related kidney disease (lupus nephritis - LN), or anti-neutrophil cytoplasmic antibody (ANCA) associated vasculitis (AAV) to determine if povetacicept is safe and potentially beneficial in treating these diseases.

During the study treatment period, participants will receive povetacicept approximately every 4 weeks for 6 months, with the possibility of participating in a 6-month treatment extension period and an optional 52-week treatment extension period. Participants with IgAN and pMN may also receive povetacicept for an additional 52 weeks, if eligible.

ELIGIBILITY:
Key Inclusion Criteria Summary:

Part A:

* Biopsy-confirmed autoantibody-associated glomerular disease: immunoglobulin A nephropathy (IgAN), primary membranous nephropathy (pMN), or lupus nephritis (LN)
* On maximal dose or the maximally tolerated dose ACEis/ARBs for ≥12 weeks prior to study Day 1
* Indication-specific criteria:

  1. IgAN

     * Biopsy-confirmed diagnosis less than or equal to (≤)10 years prior to the start of screening AND Screening UPCR greater than or equal to (≥)0.5 g/g.
     * No background immunosuppression therapies.
  2. pMN

     * A historical biopsy-confirmed diagnosis with positive anti-PLA2R1 antibodies or anti-THSD7A antibodies at screening AND Screening UPCR ≥1 g/g
     * Inadequate reduction of proteinuria determined by the Principal Investigator (PI) despite optimal supportive care for at least 12 weeks.
     * No background immunosuppression therapies except for optional calcineurin inhibitors.
  3. LN

     * A Biopsy-confirmed diagnosis of active, proliferative Class III, IV, (with or without Class V) LN ≤6 months prior to the start of screening AND Screening UPCR ≥1 g/g,
     * Anti-dsDNA at screening. Anti-dsDNA testing is required but the result need not be positive.
     * On stable background immunosuppression ≥ 8 weeks prior to Day 1
  4. AAV

     * Past diagnosis of renal AAV, defined as either of the following:
     * History of renal biopsy consistent with renal AAV.
     * History of clinically diagnosed renal AAV.
     * Myeloperoxidase (MPO)-ANCA or proteinase 3 (PR3)-ANCA positive by enzyme-linked immunosorbent assay at screening.
     * At least 4 weeks since initiation of AAV induction therapy, if applicable.

     Part B:
* Participants meet at least 1 of the following criteria:

  * Completed investigational product (IP) treatment and 24 weeks of follow-up in Part A, or
  * Had IP interruption(s) in Part A, but did not permanently discontinue IP, and completed study visits up to the last scheduled visit of the follow-up period of Part A.

Key Exclusion Criteria Summary:

Part A:

* Prior diagnosis of, or fulfills diagnostic criteria for, another renal disease
* eGFR <30 milliliter per minute per square meter (mL/min/1.73m^2) or rapidly progressive glomerulonephritis
* Recent serious or ongoing infection; risk or history of serious infection
* Receipt of B cell depleting therapies or anti-BAFF and/or APRIL therapies within protocol specified timeframes

Part B:

* History of poor compliance with IP and/or procedures in Part A, as deemed by the investigator or Sponsor
* History of any AEs or clinical conditions during Part A or emerging thereafter that may pose a safety concern for participation in Part B as deemed by investigator or Sponsor.

Other protocol defined Inclusion/Exclusion criteria will apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2028-03-02 (Estimated); Study Completion 2028-03-02 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Study Day 1 Through 24 Weeks After Last Dose Of Study Drug
Part B: Safety as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Study Day 1 Through 12 Weeks After Last Dose Of Study Drug

SECONDARY OUTCOMES:
Part A: Incidence and Titer of Anti-drug Antibodies (ADA) Against Povetacicept | Study Day 1 Through 24 Weeks After Last Dose Of Study Drug
Part B: Incidence and Titer of Anti-drug Antibodies (ADA) Against Povetacicept | Study Day 1 Through 12 Weeks After Last Dose Of Study Drug
Part A: Time Required for Povetacicept To Reach Half its Concentration (t1/2) | Study Day 1 Through 24 Weeks After Last Dose Of Study Drug
Part B: Time Required for Povetacicept To Reach Half its Concentration (t1/2) | Study Day 1 Through 12 Weeks After Last Dose Of Study Drug
Part A: Change from Baseline in Serum Ig Isotypes (IgM, total IgA, IgA1, IgA2, total IgG, IgG1, IgG2, IgG3, IgG4, IgE). | Study Day 1 Through 24 Weeks After Last Dose Of Study Drug
Part B: Change from Baseline in Serum Ig Isotypes (IgM, total IgA, IgA1, IgA2, total IgG, IgG1, IgG2, IgG3, IgG4, IgE) | Study Day 1 Through 12 Weeks After Last Dose Of Study Drug
Part A: Change from Baseline in Peripheral Blood Lymphocytes and Subsets | Study Day 1 Through 24 Weeks After Last Dose Of Study Drug
Part B: Change from Baseline in Peripheral Blood Lymphocytes and Subsets | Study Day 1 Through 12 Weeks After Last Dose Of Study Drug
Part A:Change from Baseline Over Time In Circulating Levels Of anti-dsDNA in LN; galactose deficient IgA1 (Gd-IgA1) and anti-Gd-IgA1 in IgAN; anti-PLA2R1 or anti THSD7A in pMN and anti-PR3 or anti-MPO in AAV | Study Day 1 Through 24 Weeks After Last Dose Of Study Drug
Part B: Change from Baseline Over Time In Circulating Levels Of galactose deficient IgA1 (Gd-IgA1) and anti-Gd-IgA1 in IgAN; anti-PLA2R1 or anti THSD7A in pMN | Study Day 1 Through 12 Weeks After Last Dose Of Study Drug
Part A: Change From Baseline Over Time In Complement Components (C3, C4, CH50) | Study Day 1 Through 24 Weeks After Last Dose Of Study Drug
Part B: Change From Baseline Over Time In Complement Components (C3, C4, CH50) | Study Day 1 Through 12 Weeks After Last Dose Of Study Drug
Part A: Immunological Remission (pMN only) | Study Day 1 Through Week 24 After Dose of Study Drug
Part B: Immunological Remission (pMN only) | Study Day 1 Through Week 12 After Dose of Study Drug
Part A: Change from Baseline at Week 24 in UPCR (Urine protein/creatinine ratio) (based on assessment of 24-hour urine) | Baseline and at Week 24
Part A: Change from Baseline at Week 24 in Estimated Glomerular Filtration Rate (eGFR) | Baseline and at Week 24
Part B: Change from Baseline at Week 24 in Estimated Glomerular Filtration Rate (eGFR) | Baseline and at Week 24
Part A: Renal Response | At Week 24
Part A: Remission of Vasculitis (Birmingham Vasculitis Activity Score (BVAS = 0)) (for AAV cohorts only) | At Week 24
Part A: Changes in Biomarkers Including Cytokines and Autoantibodies After Treatment with Povetacicept | Study Day 1 Through 24 Weeks After Last Dose Of Study Drug
Part B: Changes in Biomarkers Including Cytokines and Autoantibodies After Treatment with Povetacicept | Study Day 1 Through 12 Weeks After Last Dose Of Study Drug

CONTACTS AND LOCATIONS:
Locations (30):
- United States (18):
  - Investigational Site (523), Phoenix, Arizona
  - Investigational Site (501), Phoenix, Arizona
  - Investigational Site (524), Tucson, Arizona
  - Investigational Site (506), Valencia, California
  - Investigational Site (513), Arvada, Colorado
  - Investigational Site (512), Orlando, Florida
  - Investigational Site (525), Tamarac, Florida
  - Investigational Site (502), Lawrenceville, Georgia
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Investigational Site (503), Boston, Massachusetts
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Investigational Site (509), Newark, New Jersey
  - Investigational Site (511), Albany, New York
  - Investigational Site (508), Brooklyn, New York
  - Investigational Site (518), Bethlehem, Pennsylvania
  - Investigational Site (118), Colleyville, Texas
  - Investigational Site (516), Houston, Texas
  - Investigational Site (526), Irving, Texas
- Australia (3):
  - Investigational Site (519), Concord, New South Wales
  - Investigational Site (515), Saint Albans, Victoria
  - Investigational Site (102), Nedlands, Western Australia
- Investigational Site (191), Caguas, Puerto Rico
- South Korea (8):
  - Investigational Site (507), Cheonan, Chungcheongnam-do
  - Investigational Site (505), Anyang-si, Gyeonggi-do
  - Investigational Site (504), Goyang-si, Gyeonggi-do
  - Investigational Site (510), Guri-si, Gyeonggi-do
  - Investigational Site (125), Seoul, Gyeonggi-do
  - Investigational Site (520), Seoul, Gyeonggi-do
  - Investigational Site (521), Seoul, Gyeonggi-do
  - Investigational Site (116), Suwon, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing